CLINICAL TRIAL: NCT05342584
Title: Phase 1B Study of Venetoclax in Combination With Standard Intensive Chemotherapy With Daunorubicin Plus Cytarabine Followed by High-Dose Cytarabine in Adult Patients With Newly Diagnosed Acute Myeloid Leukemia and Advanced Myelodysplastic Syndrome
Brief Title: Venetoclax Plus Intensive Chemotherapy in AML and Advanced MDS
Acronym: Venetoclax AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: AbbVie (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13643
Record Dates: First submitted 2022-04-19; First posted 2022-04-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS; Venetoclax; Ven; 7+3; daunorubicin and cytarabine; daunorubicin; cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — venetoclax; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax plus 7+3 (Experimental): see detailed description
  Interventions: Drug: Venetoclax Oral Tablet; Drug: Daunorubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax Oral Tablet — Given PO
Drug: Daunorubicin — Given IV
Drug: Cytarabine — Given IV

SUMMARY:
This is a Phase 1b, open-label study evaluating Venetoclax in combination with intensive induction and consolidation chemotherapy in previously untreated, adult patients with acute myeloid leukemia. In Part 1, the dose escalation phase, the safety and tolerability of the combination with Venetoclax at different doses and duration will inform the appropriate dose(s) and regimen(s) for Part 2. In Part 2, the dose expansion phase, a maximum of 28 additional patients will be randomized 1:1 to the MTD determined in Part 1 and the starting dose (assuming the MTD is not the starting dose), to further evaluate the safety and efficacy of the study drug combination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability and determine the dose-limiting toxicity and the maximum tolerated dose (MTD) of the combination of daunorubicin & cytarabine chemotherapy plus Venetoclax for patients with AML

SECONDARY OBJECTIVES:

I. To assess efficacy by response per 2022 ELN and revised International Working Group (IWG) criteria.

II. To determine additional response parameters: CR/CRi and CR/CRh rates.

III. To determine time to response variables including overall survival (OS), event-free survival (EFS) and duration of response (DOR)

EXPLORATORY OBJECTIVES:

I. To assess MRD eradication by targeted duplex sequencing

II. To assess rates of LSC eradication by means of MFC and single cell sequencing, as well as a novel assay that uses an extended leukemia-specific NGS panel for measuring MRD in cfDNA and BM ("high resolution MRD assay")

III. To comprehensively analyze the clonal architectural and transcriptomic shifts in residual LSC under therapy

IV. To determine the protein expression of BCL-2 family members and the reliance of leukemic cells on differing members of the BH3 family at the time of diagnosis and relapse and explore association of such observations with response to Venetoclax when combined with chemotherapy

Induction Phase

Dose Escalation Cohorts:

A minimum of 3 patients will be treated in each cohort (dose level) sequentially in a 3+3 design. Patients will receive the Venetoclax plus daunorubicin/cytarabine combination as shown below

Patients aged ≤ 60 years

Cohort 1A:

Daunorubicin 60mg/m2 intravenously (IV) daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-8

Cohort 2A:

Daunorubicin 90mg/m2 IV daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-8

Cohort 3A:

Daunorubicin 60mg/m2 IV daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-11

Cohort 4A:

Daunorubicin 60mg/m2 IV daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-14

Note: No DLTs in induction phase have been observed and Cohort 3A has completed enrollment. However, the daunorubicin dose of 90mg/m2 will not be further studied due to recently reported results of no superiority over the dose of 60mg/m2.

Patients >60 years

Cohort 1B:

Daunorubicin 60mg/m2 IV daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-8

Cohort 2B:

Daunorubicin 60mg/m2 IV daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-11

Cohort 3B:

Daunorubicin 60mg/m2 IV daily on Days 2-4; Cytarabine 100mg/m2 IV daily on Days 2-8; Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-14

Expansion Cohort(s):

A maximum of 28 additional patients aged ≤ 60 years and 28 patients >60 years will be randomized (1:1) to the MTD the starting dose (assuming the MTD is not the starting dose), to further evaluate safety and efficacy of the study drug combination and identify the optimal phase 2 dose.

A. Patients aged ≤ 60 years

Expansion Cohort 1A:

Daunorubicin 60mg/m2 intravenously (IV) daily on Days 2-4 Cytarabine 100mg/m2 IV daily on Days 2-8 Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-8

Expansion Cohort 2A:

Daunorubicin 60mg/m2 intravenously (IV) daily on Days 2-4 Cytarabine 100mg/m2 IV daily on Days 2-8 Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Days 3-14

B. Patients aged > 60 years

Expansion Cohort 1B:

Daunorubicin 60mg/m2 intravenously (IV) daily on Days 2 to 4 Cytarabine 100mg/m2 IV daily on Days 2 to 8 Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Day 3 and until Day 8

Expansion Cohort 2B:

Daunorubicin 60mg/m2 intravenously (IV) daily on Days 2 to 4 Cytarabine 100mg/m2 IV daily on Days 2 to 8 Venetoclax 100mg orally on Day 1, 200mg on Day 2, 400mg on Day 3 and until Day 14

Consolidation Phase:

Patients who achieve CRc post induction will proceed to consolidation therapy with intermediate-dose cytarabine in combination with escalating doses of Venetoclax. The 3+3 algorithm will be applied for dose escalation/de-escalation of Venetoclax in combination with Cytarabine. As of February 2023, there have been 2/6 hematologic DLTs in consolidation cohort 1B, therefore Venetoclax was not given in combination with intermediate-dose cytarabine during the consolidation phase, in pts >60 yrs of age, during the dose-escalation phase of the study. In addition, dose escalation of Venetoclax during consolidation in the 60-year-old or younger age-group before RP2D of induction is determined will not be explored. All subjects ≤ 60yrs will be treated at the consolidation Cohort 1A dose.

In the expansion phase, Venetoclax, at the dose of 200mg daily, will be re-introduced in combination with chemotherapy, albeit at a shorter than a 7-day duration; the consolidation regimen for patients older than 60 years of age will consist of cytarabine at the dose of 0.5-1g/m2 every 12 hours on days 1, 3, 5 or days 1, 2, 3 (per ELN 2022 guidelines) plus Venetoclax 200mg for 5 days.

Patients ≤ 60 years

Consolidation cohort 1A:

Cytarabine 1-1.5g/m2 every 12 hours on Days 1, 3, 5 OR days 1, 2, 3; Venetoclax 200mg on Days 1-7

Patients >60 years

Consolidation cohort 1B:

Cytarabine 0.5-1g/m2 every 12 hours on days 1, 3, 5 OR days 1, 2, 3; Venetoclax 200mg on Days 1-5

A minimum of 3 patients will be treated in each cohort (dose level) sequentially in a 3+3 design. Additional 3 subjects may be backfilled to lower dose levels so that each cohort will reach a total of 6 subjects. Once the MTD is reached, a maximum of 28 additional patients will be randomized 1:1 to the MTD or a dose level below the MTD the starting dose (assuming the MTD is not the starting dose) for a total of up to 20 patients (6 from Part 1, 20 from Part 2) treated at each of those dose levels. A maximum of 52 patients (including backfill and expansion cohorts) 60 years or younger and 46 patients older than 60 years may be enrolled in this Phase 1b study.

Patients will receive 1-2 cycles of induction chemotherapy as described above. No dose adjustment of daunorubicin or cytarabine will be allowed during first induction, but may be required in second induction as described in the dose adjustment guidelines for renal insufficiency or liver dysfunction in the study protocol. Patients who do not achieve CR/CRi after a second induction will be taken off protocol and will be treated per treating physician's discretion. Patients who achieve CRc will proceed to consolidation therapy with intermediate-dose cytarabine in combination with escalating doses of Venetoclax (200-400mg) for up to four 28(-42)-day cycles, as described above (complete dose adjustment guidelines are outlined in the study protocol); consolidation with allogeneic transplantation off protocol is allowed per physician's discretion. The 3+3 algorithm will be applied for dose escalation/de-escalation of Venetoclax in combination with intermediate-dose cytarabine.

All participants should undergo response evaluations between Day 28 and Day 42 of first and/or second induction course. Unless there is clear evidence of progressive disease in the blood, bone marrow aspiration is required and bone marrow biopsy is strongly encouraged. In cases with hypocellular marrows (<10% cellularity), repeat bone marrow examinations should be considered when there is evidence of hematopoietic recovery. If multiple bone marrow examinations are performed, the last examination will be used to classify the patient's response. The final response will be determined no later than day 42 from the start of therapy.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of AML by WHO criteria. Patients with higher risk MDS (R-IPSS>3.5) and 10% blasts or more, or proliferative (WBC ≥ 13 x 10⁹/L) CMML-2 are also eligible at the discretion of the PI. Patients having received any prior hypomethylating agent with or without BCL2 inhibitor therapy for MDS/AML are also eligible at the discretion of the PI
* Patients ≥ 18 to ≤ 75 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Adequate renal function including creatinine clearance > 30 mL/min based on the Cockcroft Gault equation.
* Adequate hepatic function including total bilirubin < 1.5x ULN unless increase is due to Gilbert's disease or leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement
* Ability to understand and provide signed informed consent
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug.

Exclusion Criteria:

* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (FAB class M3-AML)
* Subject has known active CNS involvement with AML
* Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <45% by echocardiogram or multi-gated acquisition (MUGA) scan
* Patients with a history of myocardial infarction within the last 6 months or unstable / uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias
* Patients with uncontrolled infection with human immunodeficiency virus (HIV) or active Hepatitis B or C
* Patients with known dysphagia, short-gut syndrome, or other conditions that would affect the ingestion or gastrointestinal absorption of drugs administered orally.
* Subject has any other significant medical or psychiatric history that in the opinion of the investigator would adversely affect participation in this study.
* Subject has a white blood cell count > 25 x 10⁹/L. (Note: Hydroxyurea and/or cytarabine (up to 2 g/m^2 is permitted to meet this criterion.)
* Nursing women, women of childbearing potential (WOCBP) with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception. Appropriate method(s) of contraception include oral or injectable hormonal birth control, IUD, and double barrier methods (for example a condom in combination with a spermicide).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity of all Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, up to 6 years
  The number and percentage of patients with SAEs and AEs, including AEs leading to dose modifications or discontinuations, will be summarized.
Frequency and Severity of AEs and SAEs by Age Group | Through study completion, up to 6 years
  The number and percentage of patients with SAEs and AEs, including AEs leading to dose modifications or discontinuations, will be summarized by age group.
Frequency and Severity of AEs and SAEs by Dose Level | Through study completion, up to 6 years
  The number and percentage of patients with SAEs and AEs, including AEs leading to dose modifications or discontinuations, will be summarized by dose level.
Rate of Non-Hematologic Dose Limiting Toxicities (DLTs) | Up to 28 days during induction and 1st consolidation cycle
  The rate of non-hematologic DLTs will be monitored. Non-hematologic DLTs will be defined as any Grade 3 or higher non-hematologic events occurring during the first cycle (i.e., the first 28 days) that are at least possibly attributable to Venetoclax unless the event is clearly due to extraneous causes or disease progression, confirmed Hy's law case, with the exceptions outlined in Section 4.5.1 of the study protocol. The number/percentage of patients non-hematologic DLTs will be summarized. 90% Confidence Intervals will be estimated using the Clopper-Pearson method with all available data at the Maximum Tolerated Dose (MTD) and, if relevant, for the dose level below.
Rate of Hematologic Dose Limiting Toxicities (DLTs) | Up to 42 days during induction and 1st consolidation cycle
  The rate of hematologic DLTs will be monitored. Hematologic DLT is defined as Grade ≥ 3 neutropenia and/or thrombocytopenia with no greater than 5% marrow blasts lasting for 6 weeks or more after the start of a course unless the delay in count recovery is due to another identifiable factor, such as documented myelosuppressive infection. Anemia will not be considered for the definition of DLT. The number/percentage of patients with hematologic DLTs will be summarized. 90% Confidence Intervals will be estimated using the Clopper-Pearson method with all available data at the MTD and, if relevant, for the dose level below.
The Number/Percentage of Patients with Dose Modifications | During the 3 days of chemotherapy administration
  The number/percentage of patients with dose modifications, as prescribed in the protocol for the 400mg and 200mg dosage, will be summarized. It should be noted that the only relevant dose modifications apply to consolidation cycles with intermediate dose cytarabine and specifically the older group cohort.
Maximum tolerated dose of Venetoclax in combination with Daunorubicin and Cytarabine | During induction phase, up to 14 days
  To determine a safe and tolerable dose of Venetoclax in combination with Daunorubicin and Cytarabine during the induction phase.
Maximum tolerated dose of Venetoclax in combination with high dose Cytarabine | During consolidation phase, up to 7 days
  To determine a safe and tolerable dose of Venetoclax in combination high dose of Cytarabine during the consolidation phase.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Through study completion, up to 6 years
  ORR is defined as the number/percentage of patients who achieve a complete response (CR), complete response with incomplete count recovery (CRi), or partial response (PR) to treatment. ORR will be summarized by the formula: complete response (CR) + CR with incomplete blood count recovery (CRi) + partial response (PR). The number/percentage of patients will be summarized along with the 95% credible interval.
Hematologic response rate | Through study completion, up to 6 years
  Hematologic Response rate will be defined by the number/percentage of participants demonstrating improvement in hematologic parameters that do not meet criteria for Partial Response (PR) (i.e., transfusion independence and /or decline in incidence of febrile neutropenia and related hospitalizations) based on the 2022 ELN recommendations and revised IWG response criteria for AML. The number/percentage of patients will be summarized along with a 95% confidence interval.
Duration of response (DoR) | From the date of initial response, assessed up to 6 years
  DoR is defined as the number of days from the date of initial response (CRi or better) to the date of first documented disease progression/relapse or death, whichever occurs first. DoR will be calculated for all patients.
Overall survival (OS) | Through study completion, up to 6 years
  OS is defined as the duration of time from treatment initiation until a patient's death from any cause. OS will be estimated using Kaplan-Meier methods.
Event-free survival (EFS) | Through study completion, up to 6 years
  EFS is defined as the number of days from the date of treatment initiation (i.e., course 1 day 1) to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first. EFS will be calculated for all patients. In the event that neither disease progression nor death is documented prior to study termination, analysis cutoff, or the start of confounding anticancer therapy, these endpoints will be censored at the date of last tumor assessment date. EFS will be estimated using Kaplan-Meier methods.
Morphologic leukemia-free state (MLFS) | Through study completion, up to 6 years
  MLFS is the duration of time that patients maintain a state of remission based on specific bone marrow and blood criteria. For this study it will be defined as the patient having a morphologic leukemia-free state of CRMRD-, CRiMRD-, CRhMRD- without minimal residual disease. MLFS will be calculated using Kaplan-Meier methods along with the 95% confidence interval.

OTHER OUTCOMES:
Rate of LSC eradication (exploratory objective) | Through study completion, up to 6 years
  The depth of remission will be evaluated with exploratory analyses of LSC MRD negativity by flow cytometry and single cell sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Mantzaris, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Einstein Cancer Center and Children's Hospital at Montefiore (CHAM), The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mantzaris I, Goldfinger M, Uriel M, Shastri A, Shah N, Gritsman K, Kornblum NS, Shapiro L, Sica RA, Munoz A, Chambers N, Dhawan A, Verceles JA, Fehn K, Tirone B, Shah L, Clark S, Zhang C, Kim M, Cooper DL, Verma A, Konopleva M, Feldman EJ. Venetoclax plus daunorubicin and cytarabine for newly diagnosed acute myeloid leukemia: results of a phase 1b study. Blood. 2025 Apr 24;145(17):1870-1875. doi: 10.1182/blood.2024026700. PMID 39919267